CLINICAL TRIAL: NCT05734794
Title: Study of Rituximab Monotherapy VS Steroid Therapy on Children With New-onset Nephrotic Syndrome: A Randomized Controlled Trial
Brief Title: Study of Rituximab Monotherapy on Children With New-onset Nephrotic Syndrome: A Randomized Controlled Trial
Acronym: STORM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Mao Jianhua, Associate Dean, The Children's Hospital of Zhejiang University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STORM
Record Dates: First submitted 2022-11-20; First posted 2023-02-21 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Nephrotic Syndrome in Children; Rituximab
Keywords: Rituximab; Glucocorticosteroids
MeSH Terms: interventions — Rituximab; Steroids

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rituximab Group (Experimental): Rituximab dose: 4 doses of 375 mg/m2 rituximab at 1-week intervals( within +7 days).
  Interventions: Drug: Rituximab
- Steroid Group (Active Comparator): Daily oral prednisone/prednisolone 2 mg/kg/d (maximum 60 mg/d) for 6 weeks followed by alternate day prednisone/prednisolone, 1.5 mg/kg (maximum of 50 mg), for other 6 weeks.
  Interventions: Drug: Steroid

INTERVENTIONS:
Drug: Rituximab — Rituximab dose: 4 doses of 375 mg/m2 rituximab at 1-week intervals( within +7 days), associated with trimethoprim-sulfamethoxazole(25-50 mg/kg/day orally twice per day, 3 days per week. If the patient is not allergic) for three months from the first rituximab dosing date(Day 1). Four doses of rituximab are necessary whether the patient achieves complete remission.
  Arms: Rituximab Group
Drug: Steroid — Daily oral prednisone/prednisolone 2 mg/kg/d (maximum 60 mg/d) for 6 weeks followed by alternate day prednisone/prednisolone, 1.5 mg/kg (maximum of 50 mg), for other 6 weeks. Vitamin D and calcium(adjusted according to the blood calcium level) were administered for three months.
  Arms: Steroid Group

SUMMARY:
The main objective is to evaluate the effectiveness of Rituximab monotherapy versus steroid therapy on children with new-onset nephrotic syndrome within the 52-week follow-up.

DETAILED DESCRIPTION:
Nephrotic syndrome(NS) -------the most common glomerular disease in children. Steroid, as the mainstream therapy for decades, many patients suffer from adverse effects of it, such as growth impacted, fat, and glaucoma.There is a urgent need for Steroid-sparing therapy. Rituximab, as a chemical monoclonal antibody against the cluster of differentiation antigen 20(CD20), has proved to be effective in patients with frequent-relapse/steroid-dependent NS. It has also been reported to be effective in six adult patients with new-onset NS. Rituximab mono-therapy in new-onset pediatric NS patients is still unclear.

ELIGIBILITY:
Inclusion Criteria:

1. New-onset idiopathic nephrotic syndrome
2. Glomerular filtration rate (eGFR) ≥90 ml/min per 1.73 m2 at study entry.

Exclusion Criteria:

1. Glomerular hematuria: Urine red blood cell counts≥ 10/high power field(HP), ≥ 3 times within 2 weeks;
2. Continuous hypocomplementaemia(< 0.9g/L) ;
3. Repeated or persistent Hypertension(systolic and/or diastolic blood pressures measured greater than the 95th percent of blood pressure in children matching sex, age and height ≥3 different time points)
4. Diagnosis of secondary NS, such as secondary to Systemic Lupus Erythematosus, Immunoglobulin A Vasculitis(IgAV), diabetes, Hepatitis B virus(HBV) infection, etc.
5. Complicated with other kidney diseases, such as multiple renal cysts, ANCA vasculitis, urinary system abnormalities, etc;
6. With a family history of nephrotic syndrome, chronic glomerulonephritis, uremia, or other kidney diseases;
7. Other monogenic genetic diseases known as the effect the condition of nephrotic syndromes, such as Wilms' tumor 1(WT1), NPHS2, LAMB2, PLCE1, etc.
8. Congenital or acquired immunodeficiency, or patients with active tuberculosis, active Epstein-Barr virus and cytomegalovirus(CMV), acute hepatitis B, hepatitis C, HIV infection, deep fungal infection or other active infections.
9. Laboratory indicators were abnormal, such as moderate or severe neutropenia(≤1000/μL)， moderate or severe anemia(hemoglobin<9.0g/dL), Thrombocytopenia (platelet count<100* 10^12/L) or with abnormal hepatic function (Alaninetransaminase(ALT), aspartate Aminotransferase(AST) or bilirubin >2.5*upper limit of normal value and continue to increase for 2 weeks);
10. Steroid or immunosuppressive medicine for other diseases within 3 months, such as cyclophosphamide, cyclosporine, tacrolimus, mycophenolate mofetil, tripterygium wilfordii, etc.
11. With tumor, severe cardiac failure, severe hepatologic diseases, hematological diseases, or other severe system diseases.
12. Patients who are known to be allergic to rituximab;
13. History of transplantation, excluding cornea or hair transplantation;
14. The attenuated live vaccine was inoculated within 1 month before enrollment;
15. Patients who participated in other clinical trials within three months before enrollment;
16. Patients are not suitable for inclusion in the trial by any investigator.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2023-02-09 (Actual); Primary Completion 2025-12-25 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival time(day) after first complete remission | From complete remission to 52 weeks
  The time from complete remission to the first relapse during the whole 52-week follow-up in patients who achieve complete remission within 6 weeks. In order to evaluate the remission, all the participants will document their proteinuria. Relapse is defined by first-morning urine dipstick ≥3+ on three or more consecutive days, 24-h PCR≥2.0g/g, or 24-h urine protein ≥ 50mg/kg, with or without edema after complete remission(KDIGO 2021 Clinical Practice Guideline for the Management of Glomerular Diseases). Complete remission is defined by the first morning or 24h PCR ≤ 0.2g/g (or negative or trace dipstick) on three or more consecutive occasions(KDIGO 2021 Clinical Practice Guideline for the Management of Glomerular Diseases).

SECONDARY OUTCOMES:
Complete remission of nephrotic syndrome | From admission day to 6 weeks
  Complete remission is defined by the first morning or 24h PCR ≤ 0.2g/g (or negative or trace dipstick) on three or more consecutive occasions (KDIGO 2021 Clinical Practice Guideline for the Management of Glomerular Diseases). It will be recorded as "1" when patients achieve complete remission, or as "0".
Inefficiency of nephrotic syndrome | From admission day to 6 weeks
  Inefficiency is defined as patients still have nephrotic-range proteinuria(first-morning urine dipstick ≥3+dipstick, 24-h PCR≥2.0g/g, or 24-h urine protein ≥ 50mg/kg) after 6-week treatment.
The time(day) to first complete remission | From admission day to 6 weeks
  The time(day) from the first medicine administration to complete remission within 6 weeks.Complete remission is defined by the first morning or 24h PCR ≤ 0.2g/g (or negative or trace dipstick) on three or more consecutive occasions (KDIGO 2021 Clinical Practice Guideline for the Management of Glomerular Diseases).
Relapse of nephrotic syndrome | From admission day to 52 weeks
  Relapse is defined as patients who have first-morning urine dipstick ≥3+ on three or more consecutive days, 24-h PCR≥2.0g/g, or 24-h urine protein ≥ 50mg/kg, with or without edema after complete remission(KDIGO 2021 Clinical Practice Guideline for the Management of Glomerular Diseases). It will be recorded as "1" when patients have a relapse, or as "0".
Cumulative prednisone dosage of each individual (milligrams per kilogram per year) | From admission day to 52 weeks
  The total dosage of prednisone for each individual from the beginning to the end of the trial.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Veltkamp F, Rensma LR, Bouts AHM; LEARNS consortium. Incidence and Relapse of Idiopathic Nephrotic Syndrome: Meta-analysis. Pediatrics. 2021 Jul;148(1):e2020029249. doi: 10.1542/peds.2020-029249. Epub 2021 Jun 30. PMID 34193618
- [Background] Eddy AA, Symons JM. Nephrotic syndrome in childhood. Lancet. 2003 Aug 23;362(9384):629-39. doi: 10.1016/S0140-6736(03)14184-0. PMID 12944064
- [Background] Filler G, Young E, Geier P, Carpenter B, Drukker A, Feber J. Is there really an increase in non-minimal change nephrotic syndrome in children? Am J Kidney Dis. 2003 Dec;42(6):1107-13. doi: 10.1053/j.ajkd.2003.08.010. PMID 14655180
- [Background] Tarshish P, Tobin JN, Bernstein J, Edelmann CM Jr. Prognostic significance of the early course of minimal change nephrotic syndrome: report of the International Study of Kidney Disease in Children. J Am Soc Nephrol. 1997 May;8(5):769-76. doi: 10.1681/ASN.V85769. PMID 9176846
- [Background] Noone DG, Iijima K, Parekh R. Idiopathic nephrotic syndrome in children. Lancet. 2018 Jul 7;392(10141):61-74. doi: 10.1016/S0140-6736(18)30536-1. Epub 2018 Jun 14. PMID 29910038
- [Background] Ye Q, Mao JH. [Immunologic pathogenesis of idiopathic nephrotic syndrome in children: the present and future]. Zhonghua Er Ke Za Zhi. 2020 Sep 2;58(9):705-707. doi: 10.3760/cma.j.cn112140-20200626-00664. Chinese. PMID 32872709
- [Background] Iijima K, Sako M, Nozu K. Rituximab for nephrotic syndrome in children. Clin Exp Nephrol. 2017 Apr;21(2):193-202. doi: 10.1007/s10157-016-1313-5. Epub 2016 Jul 15. PMID 27422620
- [Background] Sinha A, Bagga A. Rituximab therapy in nephrotic syndrome: implications for patients' management. Nat Rev Nephrol. 2013 Mar;9(3):154-69. doi: 10.1038/nrneph.2012.289. Epub 2013 Jan 22. PMID 23338210
- [Background] Ravani P, Ponticelli A, Siciliano C, Fornoni A, Magnasco A, Sica F, Bodria M, Caridi G, Wei C, Belingheri M, Ghio L, Merscher-Gomez S, Edefonti A, Pasini A, Montini G, Murtas C, Wang X, Muruve D, Vaglio A, Martorana D, Pani A, Scolari F, Reiser J, Ghiggeri GM. Rituximab is a safe and effective long-term treatment for children with steroid and calcineurin inhibitor-dependent idiopathic nephrotic syndrome. Kidney Int. 2013 Nov;84(5):1025-33. doi: 10.1038/ki.2013.211. Epub 2013 Jun 5. PMID 23739238
- [Background] Chan EY, Yu ELM, Angeletti A, Arslan Z, Basu B, Boyer O, Chan CY, Colucci M, Dorval G, Dossier C, Drovandi S, Ghiggeri GM, Gipson DS, Hamada R, Hogan J, Ishikura K, Kamei K, Kemper MJ, Ma AL, Parekh RS, Radhakrishnan S, Saini P, Shen Q, Sinha R, Subun C, Teo S, Vivarelli M, Webb H, Xu H, Yap HK, Tullus K. Long-Term Efficacy and Safety of Repeated Rituximab to Maintain Remission in Idiopathic Childhood Nephrotic Syndrome: An International Study. J Am Soc Nephrol. 2022 Jun;33(6):1193-1207. doi: 10.1681/ASN.2021111472. Epub 2022 Mar 30. PMID 35354600
- [Background] Fenoglio R, Sciascia S, Beltrame G, Mesiano P, Ferro M, Quattrocchio G, Menegatti E, Roccatello D. Rituximab as a front-line therapy for adult-onset minimal change disease with nephrotic syndrome. Oncotarget. 2018 Jun 22;9(48):28799-28804. doi: 10.18632/oncotarget.25612. eCollection 2018 Jun 22. PMID 29989000